CLINICAL TRIAL: NCT07379762
Title: Comparison of Intramuscular Versus Rectal Diclofenac Sodium in Post Caesarean Pain Relief
Brief Title: Intramuscular Versus Rectal Diclofenac for Pain Relief After Cesarean Section in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CMH Multan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Rimsha Irshad, Principal Investigator, CMH Multan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1334-5132
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section Pain; Diclofenac; Suppository; Postoperative Pain
Keywords: cesarean section; postoperative pain; Diclofenac suppository; Diclofenac intramuscular
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IM Diclo (Experimental): Intramuscular diclofenac will be given for first 24-hours
  Interventions: Drug: Diclofenac 75mg
- Rectal Diclo (Active Comparator): Diclofenac suppository will be given after caesarean section for first 24-hours
  Interventions: Drug: Diclofenac 50mg

INTERVENTIONS:
Drug: Diclofenac 75mg — Participants will be given intramuscular diclofenac 75mg 8hourly for first 24-hours after cesarean section
  Other Names: Diclofenac sodium; Voltarol
  Arms: IM Diclo
Drug: Diclofenac 50mg — Participants will be given diclofenac suppository every 8 hours for first 24-hours after cesarean section
  Arms: Rectal Diclo

SUMMARY:
The goal of this clinical study is to find out which way of giving diclofenac sodium provides better pain relief after a planned cesarean section: an injection into the muscle or a suppository given through the rectum. Diclofenac is a commonly used pain-relieving medicine after surgery.

Women often experience moderate pain after a cesarean section, and effective pain control helps with early movement, breastfeeding, and overall recovery. Different methods of giving the same medicine may work differently and may affect how comfortable patients feel after surgery. This study compares these two methods to see which one reduces pain more effectively.

Researchers will compare post-operative pain levels in women who receive intramuscular diclofenac with those who receive rectal diclofenac after elective cesarean section.

The main questions this study aims to answer are:

* Does intramuscular diclofenac provide better pain relief than rectal diclofenac after cesarean section?
* Is there a difference in the need for additional (rescue) pain medicine between the two groups?

Participants will be women aged 20 to 45 years who are undergoing a planned cesarean section at term. A total of 60 women will take part in the study. They will be randomly assigned to one of two groups:

* One group will receive diclofenac as an intramuscular injection every 8 hours for the first 24 hours after surgery.
* The other group will receive diclofenac as a rectal suppository every 8 hours for the same period.

All participants will receive standard spinal anesthesia for surgery. Pain will be measured using a simple pain scale at 1, 6, 12, and 24 hours after the operation. If a participant reports significant pain, additional pain medicine will be given.

The results of this study will help doctors choose the most effective and comfortable method of pain relief for women after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 37 - 42 weeks of gestation
* planned to go for elective cesarean section

Exclusion Criteria:

* Women already on long-term analgesics
* known hypersensitivity to any of the study medications
* known diabetics (chronic or GDM)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Pain will be assessed at 1, 6, 12 and 24-hours after cesarean section
  Pain will be assessed on visual analog scale by the blinded assessor

SECONDARY OUTCOMES:
Rescue Analgesia | From cesarean section to 24-hours postoperatively
  In cases of VAS > 4, extra analgesia (rescue analgesia) will be given to control pain

CONTACTS AND LOCATIONS:
Overall Officials: Nidda Y Assistant Professor, FCPS, Study Chair — CMH Multan Institute of Medical Sciences
Locations (1):
- CMH Multan Institute of Medical Sciences, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No